CLINICAL TRIAL: NCT06505226
Title: Evaluating the Impact of Community-Based Mindfulness and Musical Programs on Psychiatric Measures, Music Mindfulness Study 2a.
Brief Title: Music Mindfulness Study 2a.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000028866_a; 2R25MH071584-11 (NIH)
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Mental Health Issue; COVID-19
Keywords: Mindfulness; Meditation; Music
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Screening prior to the consent process will include assessing the age and relevant medical history of each prospective participant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In person with live music (Experimental): Cohort 1 will be guided through in-person meditation. Participants in all cohorts will be asked to attend one of the weekly sessions offered twice a week for the entirety of the 8 weeks for at least 1 hour. Participants will also be given access and asked to listen to virtual music-backed mindfulness guided meditations to listen to between in- person sessions.
  Interventions: Behavioral: in person meditation
- In person with headphones (Experimental): Cohort 2 (also in-person) will experience this same meditation as Cohort 1 concurrently through headphones (in a space separate from Cohort 1). Participants in all cohorts will be asked to attend one of the weekly sessions offered twice a week for the entirety of the 8 weeks for at least 1 hour. Participants will also be given access and asked to listen to virtual music-backed mindfulness guided meditations to listen to between in- person sessions.
  Interventions: Behavioral: in person meditation using headphones
- Virtual participation (Experimental): Cohort 3 will be participating virtually by following along to the guided meditation via a password-protected Zoom room. Participants in all cohorts will be asked to attend one of the weekly sessions offered twice a week for the entirety of the 8 weeks for at least 1 hour. Participants will also be given access and asked to listen to virtual music-backed mindfulness guided meditations to listen to between in- person sessions.
  Interventions: Behavioral: virtual meditation

INTERVENTIONS:
Behavioral: in person meditation — in person guided meditation
  Arms: In person with live music
Behavioral: in person meditation using headphones — in person meditation using headphones
  Arms: In person with headphones
Behavioral: virtual meditation — virtually guided meditation via Zoom
  Arms: Virtual participation

SUMMARY:
Mental health vulnerability due to stress is increased in People of African Descent (PADs) in America due to disproportionate effects of racism, poverty, education, and criminal justice sentencing. Various meditation and mindfulness approaches have provided evidence of measured reductions in multiple negative dimensions of stress. However, the majority of these studies do not have an adequate representation of PADs or other marginalized groups and are not designed to be culturally relevant or community based. Music has been shown to alleviate multiple symptoms of stress and has been shown to be a preferred and effective support for meditation and mindfulness. However, its role in stress management in PADs engaged in meditation or mindfulness is seldom studied. This study aims to evaluate the effects of a virtual, community-based music mindfulness program on stress management in PAD community members with anxiety and depression during COVID19.

Music Mindfulness Study: Investigators will compare the effects of music-backed guided mindfulness mediation and guided mediation alone in alleviating anxiety and depression.

DETAILED DESCRIPTION:
Investigators hypothesize that this intervention will lead to reductions in scores on stress scales and will provide preliminary data for studies evaluating these types of community programs as an adjunct to the standard of care.

Participants will be screened, consented, and enrolled into either a 2-week pilot study (to test the feasibility of the experiment) or an 8-week full length study. The focus of this registration is the 8-week full length study.

Upon completion of the study, participants will be asked to take part in a focus group that will provide valuable feedback on their experience with the mindfulness intervention.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of anxiety or depression assessed by PHQ9 (>9) and GAD7 (>9)

Exclusion Criteria:

* Component 2a
* PHQ-9 <9, GAD7 < 9
* regular meditation practice of at least once a week
* has taken meditation course or intervention in the past year
* any hospitalizations in the last 6 months
* suicidal ideation, self-injurious behavior, or homicidal ideation at screening
* active audio-visual hallucinations or other signs of psychosis
* diagnosis of a seizure disorder or other neurological disorder that precludes outpatient participation
* history of thyroid or cardiovascular disease
* current substance use disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Mean Score Perceived Stress Scale | 8 weeks
  The Perceived Stress Scale (PSS-10) is a 10-item, validated, self-report, questionnaire used to assess perceived control and confidence in managing stressful situations over the past month. Scores range from 0 to 40, with higher scores indicated higher levels of perceived stress.

SECONDARY OUTCOMES:
Mean Score Social Connectedness Scale | 8 weeks
  The Social Connectedness Scale (SCS) is a self-report questionnaire that measures the extent to which individuals feel connected to others in their social environment. 20 items on a 6-point Likert scale, from 1 (strongly disagree) to 6 (strongly agree). Total score is achieved by summing all items with total score range from 20-120. Higher scores indicate a greater sense of social connectedness.

CONTACTS AND LOCATIONS:
Overall Officials: AZA Allsop, MD, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - BLOOM, New Haven, Connecticut
  - Musical Intervention Studios, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
De-identified, aggregate data will be shared through pre-prints, publications, and community town hall meetings.